CLINICAL TRIAL: NCT05042037
Title: The Effectiveness and Tolerability of Multi-Strain Probiotics as Adjunctive Preventive Treatment of Episodic Migraine: A Single Centre, Randomised, Double- Blind, Sham-Controlled Phase 2 Trial (PROBIOTICS -EM).
Brief Title: Probiotics as Adjunctive Migraine Prophylaxis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Wan Aliaa Wan Sulaiman, Associate professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JKEUPM-2021-276
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Migraine; Episodic Migraine
Keywords: Episodic migraine, probiotics, effectiveness, preventive treatment, randomized controlled trial.
MeSH Terms: conditions — Migraine Disorders | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment involves two groups of participants. One group receives probiotics , and the other group receives placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care provider, investigator and outcome assessor of the study is blinded about the allocation status of the participants (Double blinded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-blind, placebo-controlled interventional study (Active Comparator): Active treatment group will receive a 3-gram sachet of probiotics containing multi-strain of lactobacillus and Bifidobacterium 30 Colony Forming Unit x 109 to be taken twice daily for 12 weeks.
  Interventions: Dietary Supplement: (Microbial cell preparation) probiotics
- Placebo (Placebo Comparator): Patients will be given placebo sachet (exactly the same packaging as active comparator) to be taken 1 sachet twice daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: (Microbial cell preparation) probiotics — Lactobacillus acidophilus (107mg), Lactobacillus casei subsp (107mg), Lactobacillus lactis (107mg), Bifidobacterium bifidum (107mg), Bifidobacterium infantis (107mg) and Bifidobacterium longum (107mg)
  Other Names: Granulated Multi-strain Probiotics; Hexbio
  Arms: Double-blind, placebo-controlled interventional study
Other: Placebo — Placebo sachet with no microbial cell preparation
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of multi-strain probiotics as an adjunctive treatment for episodic migraine

DETAILED DESCRIPTION:
This is a phase 2 and single center, randomized, placebo-controlled double-blind clinical Trial. Episodic migraine patients according to International Headache Society criteria will be allocated randomly into two treatment arms. One group will receive active probiotics and another group will receive placebo for treatment phase. Both groups of patients will consume the treatment twice daily for 12 weeks and assessment will be made at baseline, baseline, week 4, 8 and 12

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fulfilling criteria for episodic migraine as per the Third Edition of The International Headache Society (ICHD-3) (Table 1)
2. Patients diagnosed with episodic migraine (4 or more episodes per month) for a minimum of 3 months.
3. On a steady treatment regimen: preventive and acute migraine medications and therapies unchanged over the last 3 months
4. Adult patients Age > 18 years old
5. A signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study including any known and potential risks and available alternative treatments.

Exclusion Criteria:

1. Lactose intolerance
2. Previous history of small and large bowel surgery
3. Use of probiotics or antibiotics in 2 weeks before baseline visit.
4. Patients with medical conditions such as severe hypertension, infections,
5. Malignancy, cardiovascular and cerebrovascular diseases, epilepsy, degenerative central nervous system diseases, renal failure, hepatic failure, bleeding diathesis and serious mental illnesses
6. Headache with red flags symptoms that may suggest organic secondary headaches.
7. Onset of headache more than 50 years
8. Prior GI infection in the previous 3-months
9. Morbid obesity (BMI >40)
10. Pregnant or lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean monthly migraine days (MMD). | Baseline, week 4, 8 and 12 post treatment
  The MMD will be calculated using the MMD recorded by patients in a headache diary from each of the months of the double-blind treatment phase.

SECONDARY OUTCOMES:
Change from baseline in mean monthly migraine attacks | Baseline, week 4, 8 and 12 post treatment
  The mean monthly migraine attacks will be calculated using the monthly migraine attack recorded by patients in headache diaries from each of the months of the double-blind treatment phase
Reduction mean monthly migraine days(MMD) | 12 weeks post treatment
  Proportion of subjects with at least a 50% reduction from baseline in MMD
Change from baseline in mean monthly pain intensity of migraine attacks | Baseline, week 4, 8 and 12 post treatment
  The mean monthly pain intensity will be based on the record of the maximal pain intensity by means of a verbal scale (i.e., 0 =no headache; 1 = mild headache; 2 = moderate headache; 3 = severe headache) prior to taking symptomatic medication
Adverse events in response to probiotics | Week 4, 8 and 12 treatment
  Frequency and adverse events in response to (probiotics)
Change from baseline in mean Migraine Induced Disability Assessment Score (MIDAS) | Week 0 and 12 post treatment
  Change from baseline in mean Migraine Induced Disability Assessment Score (MIDAS) in migraine patients in response to probiotics
Change from baseline in mean Depression, Anxiety and Stress Scale (DASS21) | Week 0 and 12 post treatment
  Change from baseline in mean Depression, Anxiety and Stress Scale (DASS21) score in migraine patients in response to probiotics
Change from baseline in mean Migraine-Specific Quality-of-Life Questionnaire (MSQ V2) score | Week 0 and 12 post treatment
  Change from baseline in mean Migraine-Specific Quality-of-Life Questionnaire (MSQ V2) score in migraine patients in response to probiotics
Serum Highly sensitive C-Reactive Protein (hs-CRP) | Week 0 and 12 post treatment
  Highly sensitive C-Reactive Protein (hs-CRP) level changes in migraine patients in response to probiotics
Serum Interleukin 6 (IL- 6) | Week 0 and 12 post treatment
  Interleukin 6 (IL- 6) level changes in migraine patients in response to probiotics
Serum Tumour Necrosis Factor Alpha (TNF-alpha) | Week 0 and 12 post treatment
  Tumour Necrosis Factor Alpha (TNF-alpha) level changes in migraine patients in response to probiotics
Satisfaction measures of efficacy, tolerability, safety, and expectations of probiotics among the participants | Week 0 and 12 post treatment
  A 5-point, Likert scale will be used to evaluate satisfaction with probiotics in migraine prevention

CONTACTS AND LOCATIONS:
Overall Officials: Hamidon Basri, AM, Study Chair — University Putra Malaysia; Wan Aliaa Wan Sulaiman, FRCP, Principal Investigator — University Putra Malaysia; Azliza Ibrahim, MMed, Study Director — Universiti Putra Malaysia
Locations (1):
- University Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No